CLINICAL TRIAL: NCT05672498
Title: A Comparative Study on the Therapeutic Effect of a Traditional Chinese Medicine Formulation on COVID-19 Infection
Brief Title: Effect of a Traditional Chinese Medicine Formulation on COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-436
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM treatment (Active Comparator): The patients are treated with traditional Chinese medicine. They take 150ml of liquid medicine every morning and evening for 7 days.
  Interventions: Drug: Traditional Chinese Medicine Formulation
- placebo treatment (Placebo Comparator): The patients are treated with placebo. They take 150ml of liquid placebo every morning and evening for 7 days .
  Interventions: Other: Placebo Treatment

INTERVENTIONS:
Drug: Traditional Chinese Medicine Formulation — The TCM Treatment Group：The patient are given a traditional Chinese medicine formulation, taking 150 ml of liquid medicine every morning and evening for 7 days.
  Arms: TCM treatment
Other: Placebo Treatment — Placebo Treatment Group:The patient are given placebo, taking 150 ml of liquid placebo every morning and evening for 7 days. All medications and placebo are packed identically in packing bags with the same labeling form.
  Arms: placebo treatment

SUMMARY:
Traditional Chinese medicine (TCM) has been handed down for thousands of years. It has a long history in the treatment of virus infection and has a good effect on the upper respiratory tract infection.

In recent years, the project applicant has been conducting research on the anti infection and anti inflammation treatment of traditional Chinese medicine, and has carried out a lot of clinical practice exploration in non-specific inflammation.

The purpose of this research is to study the therapeutic effect of a traditional Chinese medicine prescription on COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* In the past two to three days, COVID-19 test was positive, accompanied by more than one clinical symptom.
* 18 ≤ age ≤ 65, regardless of gender;
* Patients have good follow-up compliance.

Exclusion Criteria:

* Human immunodeficiency virus - 1 infection and malignant tumors; Active cardiovascular, kidney, lung, liver, blood, digestive, neurological or psychiatric diseases; Recent acute respiratory symptoms (within 4 weeks) .
* Any drug that may interfere with the evaluation (for example, other herbal products such as Lianhua Qingwen, immunosuppressants, anticoagulants), or a history of allergy or other adverse reactions to traditional Chinese medicine products.
* Pregnant or lactating women.
* Allergic constitution and allergy to multiple drugs.
* According to the judgment of the investigator, the subject suffers from any disease that may endanger his safety or affect his compliance with the protocol, or other conditions that are not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-05 (Estimated); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-05-05 (Estimated)

PRIMARY OUTCOMES:
negative Covid-19 test result | in 7 days or after the intervention
  negative test result
Disappearance or Improvement of the most common clinical symptoms | in 7 days or after the intervention
  such as fever,cough,pharyngalgia

SECONDARY OUTCOMES:
erythrocyte sedimentation rate | in 7 days or after the intervention
  mm/h
C-reactionprotein | in 7 days or after the intervention
  mg/L
Interleukin- 6 | in 7 days or after the intervention
  Pg/ml
Procalcitonin | in 7 days or after the intervention
  mg/L
Covid-19 antibody concentration | in 7 days or after the intervention
  ng/ml
blood fat | in 7 days or after the intervention
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Study Chair — First Affilicated Hospital of Xian Jiaotong University
Locations (1):
- First Affilicated Hospital of Xian Jiaotong University, Xi’an, Shanxi, China